CLINICAL TRIAL: NCT07042399
Title: Self-care Behaviours of Type 2 Diabetes Mellitus Patients: a Multicenter Prospective Observational Study With 2 Years Follow-up (SCUDOS)
Brief Title: Self-care Behaviors of Type 2 Diabetes Mellitus Patients
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Davide Ausili, Associate Professor of Nursing Science, University of Milano Bicocca
Other Study IDs: SCUDOS
Record Dates: First submitted 2023-02-16; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
Keywords: Self-care; Chronic diseases; Type 2 diabetes; Self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to explore the experience of the chronic disease, with a particular focus on self-care, in adults with type 2 diabetes mellitus. The main questions it aims to answer are:

* what is the association between self-care and glycated hemoglobin over time?
* what are participants' clinical and sociodemographic characteristics influencing self-care behaviors? Participants' socio-demographic and clinical data will be collected by medical records and, at the beginning or at the end of the clinical standard outpatient visit, they will be asked to complete study questionnaires.

The results of this study could be helpful in providing quality assistance, improving resource consumption, and reducing the onset of complications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes;
* Age over 18 years old;
* Adequate comprehension of the Italian language;
* Signed and dated informed consent.

Exclusion Criteria:

* Presence of documented psychiatric or neurodegenerative disease;
* Pregnancy;
* Any condition that, by the investigators' judgment, may limit adherence to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample will be enrolled among diabetic patients who access hospital diabetes outpatient clinics in Lombardy (a region in the North of Italy)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Self-care in diabetes [1] | The SCODI will be administered at the following time point: T0 - Baseline.
  The Self-Care of Diabetes Inventory (SCODI) is the self-report tool used to measure self-care dimensions: self-care maintenance, self-care monitoring, and self-care management.The self-care maintenance scale measures adherence to main diabetes treatments (i.e. medication, diet exercise). The self-care monitoring scale includes body listening behaviours, such as blood glucose or blood pressure monitoring and symptom recognition behaviours. The self-care management scale includes those behaviours performed by patients to manage symptoms, high or low blood glucose levels, and health problems when they occur. Furthermore, the SCODI allows to measure self-care confidence that is the degree of confidence a patient has in her/his ability to perform adequate self-care. A 5-points Likert type scale measures every item of the SCODI. All the SCODI scales provide a 0-100 standardized score where higher scores mean better self-care.
Self-care in diabetes [2] | The SCODI will be administered by telephone at the following time point: T0.5 - Month 6 ± 28 days
  The Self-Care of Diabetes Inventory (SCODI) is the self-report tool used to measure self-care dimensions: self-care maintenance, self-care monitoring, and self-care management.The self-care maintenance scale measures adherence to main diabetes treatments (i.e. medication, diet exercise). The self-care monitoring scale includes body listening behaviours, such as blood glucose or blood pressure monitoring and symptom recognition behaviours. The self-care management scale includes those behaviours performed by patients to manage symptoms, high or low blood glucose levels, and health problems when they occur. Furthermore, the SCODI allows to measure self-care confidence that is the degree of confidence a patient has in her/his ability to perform adequate self-care. A 5-points Likert type scale measures every item of the SCODI. All the SCODI scales provide a 0-100 standardized score where higher scores mean better self-care.
Self-care in diabetes [3] | The SCODI will be administered by telephone at the following time point: T1 - Month 12 ± 28 days.
  The Self-Care of Diabetes Inventory (SCODI) is the self-report tool used to measure self-care dimensions: self-care maintenance, self-care monitoring, and self-care management.The self-care maintenance scale measures adherence to main diabetes treatments (i.e. medication, diet exercise). The self-care monitoring scale includes body listening behaviours, such as blood glucose or blood pressure monitoring and symptom recognition behaviours. The self-care management scale includes those behaviours performed by patients to manage symptoms, high or low blood glucose levels, and health problems when they occur. Furthermore, the SCODI allows to measure self-care confidence that is the degree of confidence a patient has in her/his ability to perform adequate self-care. A 5-points Likert type scale measures every item of the SCODI. All the SCODI scales provide a 0-100 standardized score where higher scores mean better self-care.
Self-care in diabetes [4] | The SCODI will be administered by telephone at the following time point: T1.5 - Month 18 ± 28 days.
  The Self-Care of Diabetes Inventory (SCODI) is the self-report tool used to measure self-care dimensions: self-care maintenance, self-care monitoring, and self-care management.The self-care maintenance scale measures adherence to main diabetes treatments (i.e. medication, diet exercise). The self-care monitoring scale includes body listening behaviours, such as blood glucose or blood pressure monitoring and symptom recognition behaviours. The self-care management scale includes those behaviours performed by patients to manage symptoms, high or low blood glucose levels, and health problems when they occur. Furthermore, the SCODI allows to measure self-care confidence that is the degree of confidence a patient has in her/his ability to perform adequate self-care. A 5-points Likert type scale measures every item of the SCODI. All the SCODI scales provide a 0-100 standardized score where higher scores mean better self-care.
Self-care in diabetes [5] | The SCODI will be administered by telephone at the following time point: T2 - Month 24 ± 28 days.
  The Self-Care of Diabetes Inventory (SCODI) is the self-report tool used to measure self-care dimensions: self-care maintenance, self-care monitoring, and self-care management.The self-care maintenance scale measures adherence to main diabetes treatments (i.e. medication, diet exercise). The self-care monitoring scale includes body listening behaviours, such as blood glucose or blood pressure monitoring and symptom recognition behaviours. The self-care management scale includes those behaviours performed by patients to manage symptoms, high or low blood glucose levels, and health problems when they occur. Furthermore, the SCODI allows to measure self-care confidence that is the degree of confidence a patient has in her/his ability to perform adequate self-care. A 5-points Likert type scale measures every item of the SCODI. All the SCODI scales provide a 0-100 standardized score where higher scores mean better self-care.

SECONDARY OUTCOMES:
Glycated Hemoglobin (HbA1c) [1] | The HbA1c blood level will be collected from medical records at the following time point: T0 - Baseline.
  Blood glycated hemoglobin measured in both mmol/mol and % was used as an index of patients' glycemic control.
Glycated Hemoglobin (HbA1c) [2] | The HbA1c blood level will be collected from medical records at the following time point: T1 - Month 12± 28 days.
  Blood glycated hemoglobin measured in both mmol/mol and % was used as an index of patients' glycemic control.
Glycated Hemoglobin (HbA1c) [3] | The HbA1c blood level will be collected from medical records at the following time point: T2 - Month 24 ± 28 days.
  Blood glycated hemoglobin measured in both mmol/mol and % was used as an index of patients' glycemic control.

OTHER OUTCOMES:
Lipidic profile [1] | The lipidic profile will be collected from medical records at the following time point: T0 - Baseline.
  Blood concentration of Total Cholesterol, HDL Cholesterol, LDL Cholesterol, and Triglycerides measured in mg/dL.
Lipidic profile [2] | The lipidic profile will be collected from medical records at the following time point: T1 - Month 12 ± 28 days.
  Blood concentration of Total Cholesterol, HDL Cholesterol, LDL Cholesterol, and Triglycerides measured in mg/dL.
Lipidic profile [3] | The lipidic profile will be collected from medical records at the following time point: T2 - Month 24 ± 28 days.
  Blood concentration of Total Cholesterol, HDL Cholesterol, LDL Cholesterol, and Triglycerides measured in mg/dL.
Creatinine [1] | Creatinine blood level will be collected from medical records at the following time point: T0 - Baseline.
  Blood concentration of Creatinine measured in mg/dL.
Creatinine [2] | Creatinine blood level will be collected from medical records at the following time point: T1 - Month 12 ± 28 days.
  Blood concentration of Creatinine measured in mg/dL.
Creatinine [3] | Creatinine blood level will be collected from medical records at the following time point: T2 - Month 24 ± 28 days.
  Blood concentration of Creatinine measured in mg/dL.
Estimated Glomerular Filtration Rate (GFR) [1] | GFR will be collected from medical records at the following time point: T0 - Baseline.
  GFR estimation measured in mL/min/1.73m² from age, gender, and blood creatinine [1] using the Chronic Kidney Disease Epidemiology (CKD-EPI) 2021 formula.
Estimated Glomerular Filtration Rate (GFR) [2] | GFR will be collected from medical records at the following time point: T1 - Month 12 ± 28 days.
  GFR estimation measured in mL/min/1.73m² from age, gender, and blood creatinine [2] using the Chronic Kidney Disease Epidemiology (CKD-EPI) 2021 formula.
Estimated Glomerular Filtration Rate (GFR) [3] | GFR will be collected from medical records at the following time point: T2 - Month 24 ± 28 days.
  GFR estimation measured in mL/min/1.73m² from age, gender, and blood creatinine [3] using the Chronic Kidney Disease Epidemiology (CKD-EPI) 2021 formula.
Liver profile [1] | The liver profile will be assessed at the following time point: T0 - Baseline.
  Alanine transaminase (ALT), Aspartate transaminase (AST), and Gamma-glutamyltransferase (GGT) blood level measured in U/L.
Liver profile [2] | The liver profile will be collected from medical records at the following time point: T1 - Month 12 ± 28 days.
  Alanine transaminase (ALT), Aspartate transaminase (AST), and Gamma-glutamyltransferase (GGT) blood level measured in U/L.
Liver profile [3] | The liver profile will be collected from medical records at the following time point: T2 - Month 24 ± 28 days.
  Alanine transaminase (ALT), Aspartate transaminase (AST), and Gamma-glutamyltransferase (GGT) blood level measured in U/L.
Height | The height will be measured at following time point: T0 - Baseline.
  The height measured in meters.
Weight [1] | The weight will be measured at the following time point: T0 - Baseline.
  The weight detected on the scale during the visit and measured in kg.
Weight [2] | The weight will be collected from medical records at the following time point: T1 - Month 12 ± 28 days.
  The weight detected on the scale during the visit and measured in kg.
Weight [3] | The weight will be collected from medical records at the following time point: T2 - Month 24 ± 28 days.
  The weight detected on the scale during the visit and measured in kg.
Abdominal circumference [1] | Abdominal circumference will be measured at the following time point: T0 - Baseline
  Abdominal circumference measurement in cm.
Abdominal circumference [2] | Abdominal circumference will be collected from medical records at the following time point: T1 - Month 12 ± 28 days.
  Abdominal circumference measurement in cm.
Abdominal circumference [3] | Abdominal circumference will be collected from medical records at the following time point: T2 - Month 24 ± 28 days.
  Abdominal circumference measurement in cm.
Body Mass Index (BMI) [1] | The BMI will be estimated at the following time point: T0 - Baseline.
  The BMI measured in kg/m² from height and weight [1].
Body Mass Index (BMI) [2] | The BMI will be estimated at the following time point: T1 - Month 12 ± 28 days.
  The BMI measured in kg/m² from height and weight [2].
Body Mass Index (BMI) [3] | The BMI will be estimated at the following time point: T2 - Month 24 ± 28 days.
  The BMI measured in kg/m² from height and weight [3].
Blood pressure [1] | The blood pressure will be measured at the following time point: T0 - Baseline.
  The systolic and diastolic blood pressure measured di mmHg.
Blood pressure [2] | The blood pressure will be collected from medical records at the following time point: T1 - Month 12 ± 28 days.
  The systolic and diastolic blood pressure measured di mmHg.
Blood pressure [3] | The blood pressure will be collected from medical records at the following time point: T2 - Month 24 ± 28 days.
  The systolic and diastolic blood pressure measured di mmHg.
Pulse rate [1] | The pulse rate will be measured at the following time point: T0 - Baseline.
  The pulse rate measured in beats per minute (bpm).
Pulse rate [2] | The pulse rate will be collected from medical records at the following time point: T1 - Month 12 ± 28 days.
  The pulse rate measured in beats per minute (bpm).
Pulse rate [3] | The pulse rate will be collected from medical records at the following time point: T2 - Month 24 ± 28 days.
  The pulse rate measured in beats per minute (bpm).
Short Form 12 (SF-12) [1] | The SF-12 will be administered at the following time point: T0 - Baseline.
  The SF-12 evaluates the functional and mental well-being status. It has a 4 week retrospective span and inquires personal and social discomfort disabilities and self-description of the level of health perceived. It can be self-administered and it counts 12 items.
Short Form 12 (SF-12) [2] | The SF-12 will be administered by telephone at the following time point: T1 - Month 12 ± 28 days.
  The SF-12 evaluates the functional and mental well-being status. It has a 4 week retrospective span and inquires personal and social discomfort disabilities and self-description of the level of health perceived. It can be self-administered and it counts 12 items.
Short Form 12 (SF-12) [3] | The SF-12 will be administered by telephone at the following time point: T2 - Month 24 ± 28 days.
  The SF-12 evaluates the functional and mental well-being status. It has a 4 week retrospective span and inquires personal and social discomfort disabilities and self-description of the level of health perceived. It can be self-administered and it counts 12 items.
EuroQoL - 5 Dimensions - 3 Levels (EQ-5D-3L) [1] | The EQ-5D-3L will be administered at the following time points: T0 - Baseline.
  The EQ-5D-3L is a self-report tool, composed of 5 items of multiple questions that investigate the quality of life. Questions are about movement, hygiene, daily living activities tolerance, pain/discomfort, and anxiety/depression. A Visual Analogue Scale is included in order to assess a general health status level as perceived by patients
EuroQoL - 5 Dimensions - 3 Levels (EQ-5D-3L) [2] | The EQ-5D-3L will be administered by telephone at the following time point: T0.5 - Month 6 ± 28 days.
  The EQ-5D-3L is a self-report tool, composed of 5 items of multiple questions that investigate the quality of life. Questions are about movement, hygiene, daily living activities tolerance, pain/discomfort, and anxiety/depression. A Visual Analogue Scale is included in order to assess a general health status level as perceived by patients
EuroQoL - 5 Dimensions - 3 Levels (EQ-5D-3L) [3] | The EQ-5D-3L will be administered by telephone at the following time point: T1 - Month 12 ± 28 days.
  The EQ-5D-3L is a self-report tool, composed of 5 items of multiple questions that investigate the quality of life. Questions are about movement, hygiene, daily living activities tolerance, pain/discomfort, and anxiety/depression. A Visual Analogue Scale is included in order to assess a general health status level as perceived by patients
EQ-5D-3L [4] | The EQ-5D-3L will be administered by telephone at the following time point: T1.5 - Month 18 ± 28 days.
  The EQ-5D-3L is a self-report tool, composed of 5 items of multiple questions that investigate the quality of life. Questions are about movement, hygiene, daily living activities tolerance, pain/discomfort, and anxiety/depression. A Visual Analogue Scale is included in order to assess a general health status level as perceived by patients
EQ-5D-3L [5] | The EQ-5D-3L will be administered at the following time point: T2 - Month 24 ± 28 days.
  The EQ-5D-3L is a self-report tool, composed of 5 items of multiple questions that investigate the quality of life. Questions are about movement, hygiene, daily living activities tolerance, pain/discomfort, and anxiety/depression. A Visual Analogue Scale is included in order to assess a general health status level as perceived by patients
Problem Areas in Diabetes Questionnaire Short Form (PAID-5) [1] | The PAID-5 will be administered at the following time point: T0 - Baseline.
  The PAID-5 is composed by 5 items and it can be self-administered. It has satisfactory sensitivity and specificity for recognition of diabetes-related emotional distress. The final score is between 0 and 100 points: a score higher than 40 points has been significantly associated to development of depression and other negative psychological outcomes.
Problem Areas in Diabetes Questionnaire Short Form (PAID-5) [2] | The PAID-5 will be administered by telephone at the following time point: T1 - Month 12 ± 28 days.
  The PAID-5 is composed by 5 items and it can be self-administered. It has satisfactory sensitivity and specificity for recognition of diabetes-related emotional distress. The final score is between 0 and 100 points: a score higher than 40 points has been significantly associated to development of depression and other negative psychological outcomes.
Problem Areas in Diabetes Questionnaire Short Form (PAID-5) [3] | The PAID-5 will be administered by telephone at the following time point: T2 - Month 24 ± 28 days.
  The PAID-5 is composed by 5 items and it can be self-administered. It has satisfactory sensitivity and specificity for recognition of diabetes-related emotional distress. The final score is between 0 and 100 points: a score higher than 40 points has been significantly associated to development of depression and other negative psychological outcomes.
Pittsburgh Sleep Quality Index (PSQI) [1] | The PSQI will be administered at the following time point: T0 - Baseline.
  The Pittsburgh Sleep Quality Index is a tool for assessing sleep quality. It comprises 19 items and it is self-administered. It provides a good and reliable differentiation between normal and pathological groups, with higher scores (cut-off 5 and higher) reported by people characterised by more impaired sleep quality.
Pittsburgh Sleep Quality Index (PSQI) [2] | The PSQI will be administered by telephone at the following time point: T1 - Month 12 ± 28 days.
  The Pittsburgh Sleep Quality Index is a tool for assessing sleep quality. It comprises 19 items and it is self-administered. It provides a good and reliable differentiation between normal and pathological groups, with higher scores (cut-off 5 and higher) reported by people characterised by more impaired sleep quality.
Pittsburgh Sleep Quality Index (PSQI) [3] | The PSQI will be administered by telephone at the following time point: T2 - Month 24 ± 28 days.
  The Pittsburgh Sleep Quality Index is a tool for assessing sleep quality. It comprises 19 items and it is self-administered. It provides a good and reliable differentiation between normal and pathological groups, with higher scores (cut-off 5 and higher) reported by people characterised by more impaired sleep quality.
Events [1] | Events will be assessed at the following time point: T0 - Baseline.
  Any referral or unplanned diabetes visit, request for home care assistance, hospitalisation, access to emergency care, death, received diabetes education in the last year.
Events [2] | Events will be assessed by telephone and collected from medical records at the following time point: T1 - Month 12 ± 28 days.
  Any referral or unplanned diabetes visit, request for home care assistance, hospitalisation, access to emergency care, death, received diabetes education in the last year.
Events [3] | Events will be assessed by telephone and collected from medical records at the following time point: T2 - Month 24 ± 28 days.
  Any referral or unplanned diabetes visit, request for home care assistance, hospitalisation, access to emergency care, death, received diabetes education in the last year.

CONTACTS AND LOCATIONS:
Overall Officials: Davide LL Ausili, Study Director — Università degli Studi di Milano - Bicocca
Locations (2):
- Italy (2):
  - IRCCS Policlinico San Donato, San Donato Milanese, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Monza Brianza

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is foreseen between participating centers. The possibility of later sharing the data with other researchers for collaboration is considered. In any case, the data will be shared guaranteeing the anonymity of the individual participants so that it will be impossible to trace the subject.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Support information will be made sharable even before enrollment begins. IPD will be shared at the end of data collection for each time point. At the end of the follow-up, data will remain shareable for 5 years
Access Criteria: Being a researcher of one of the centers involved in the study

REFERENCES:
- [Background] Riegel B, Dunbar SB, Fitzsimons D, Freedland KE, Lee CS, Middleton S, Stromberg A, Vellone E, Webber DE, Jaarsma T. Self-care research: Where are we now? Where are we going? Int J Nurs Stud. 2021 Apr;116:103402. doi: 10.1016/j.ijnurstu.2019.103402. Epub 2019 Aug 23. PMID 31630807
- [Background] Riegel B, Jaarsma T, Lee CS, Stromberg A. Integrating Symptoms Into the Middle-Range Theory of Self-Care of Chronic Illness. ANS Adv Nurs Sci. 2019 Jul/Sep;42(3):206-215. doi: 10.1097/ANS.0000000000000237. PMID 30475237
- [Background] Riegel B, Jaarsma T, Stromberg A. A middle-range theory of self-care of chronic illness. ANS Adv Nurs Sci. 2012 Jul-Sep;35(3):194-204. doi: 10.1097/ANS.0b013e318261b1ba. PMID 22739426
- [Background] Powers MA, Bardsley J, Cypress M, Duker P, Funnell MM, Fischl AH, Maryniuk MD, Siminerio L, Vivian E. Diabetes Self-management Education and Support in Type 2 Diabetes: A Joint Position Statement of the American Diabetes Association, the American Association of Diabetes Educators, and the Academy of Nutrition and Dietetics. Clin Diabetes. 2016 Apr;34(2):70-80. doi: 10.2337/diaclin.34.2.70. No abstract available. PMID 27092016
- [Background] Yuan C, Lai CW, Chan LW, Chow M, Law HK, Ying M. The effect of diabetes self-management education on body weight, glycemic control, and other metabolic markers in patients with type 2 diabetes mellitus. J Diabetes Res. 2014;2014:789761. doi: 10.1155/2014/789761. Epub 2014 Jul 17. PMID 25136645
- [Background] Walker RJ, Smalls BL, Hernandez-Tejada MA, Campbell JA, Egede LE. Effect of diabetes self-efficacy on glycemic control, medication adherence, self-care behaviors, and quality of life in a predominantly low-income, minority population. Ethn Dis. 2014 Summer;24(3):349-55. PMID 25065078
- [Background] Shrivastava SR, Shrivastava PS, Ramasamy J. Role of self-care in management of diabetes mellitus. J Diabetes Metab Disord. 2013 Mar 5;12(1):14. doi: 10.1186/2251-6581-12-14. PMID 23497559
- [Background] Ausili D, Barbaranelli C, Rossi E, Rebora P, Fabrizi D, Coghi C, Luciani M, Vellone E, Di Mauro S, Riegel B. Development and psychometric testing of a theory-based tool to measure self-care in diabetes patients: the Self-Care of Diabetes Inventory. BMC Endocr Disord. 2017 Oct 16;17(1):66. doi: 10.1186/s12902-017-0218-y. PMID 29037177
- [Background] Ausili D, Rossi E, Rebora P, Luciani M, Tonoli L, Ballerini E, Androni S, Vellone E, Riegel B, Di Mauro S. Socio-demographic and clinical determinants of self-care in adults with type 2 diabetes: a multicentre observational study. Acta Diabetol. 2018 Jul;55(7):691-702. doi: 10.1007/s00592-018-1135-x. Epub 2018 Apr 5. PMID 29623431
- [Background] Sherwani SI, Khan HA, Ekhzaimy A, Masood A, Sakharkar MK. Significance of HbA1c Test in Diagnosis and Prognosis of Diabetic Patients. Biomark Insights. 2016 Jul 3;11:95-104. doi: 10.4137/BMI.S38440. eCollection 2016. PMID 27398023
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Savoia E, Fantini MP, Pandolfi PP, Dallolio L, Collina N. Assessing the construct validity of the Italian version of the EQ-5D: preliminary results from a cross-sectional study in North Italy. Health Qual Life Outcomes. 2006 Aug 10;4:47. doi: 10.1186/1477-7525-4-47. PMID 16901340
- [Background] McGuire BE, Morrison TG, Hermanns N, Skovlund S, Eldrup E, Gagliardino J, Kokoszka A, Matthews D, Pibernik-Okanovic M, Rodriguez-Saldana J, de Wit M, Snoek FJ. Short-form measures of diabetes-related emotional distress: the Problem Areas in Diabetes Scale (PAID)-5 and PAID-1. Diabetologia. 2010 Jan;53(1):66-9. doi: 10.1007/s00125-009-1559-5. Epub 2009 Oct 20. PMID 19841892
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Curcio G, Tempesta D, Scarlata S, Marzano C, Moroni F, Rossini PM, Ferrara M, De Gennaro L. Validity of the Italian version of the Pittsburgh Sleep Quality Index (PSQI). Neurol Sci. 2013 Apr;34(4):511-9. doi: 10.1007/s10072-012-1085-y. Epub 2012 Apr 13. PMID 22526760

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT07042399/Prot_SAP_000.pdf